CLINICAL TRIAL: NCT03723018
Title: Me-GC: A Randomized Controlled Trial of Meditation to Reduce Genetic Counselor Burnout and Genetic Counseling Student Stress
Brief Title: Me-GC: A Randomized Controlled Trial of Meditation for Genetic Counselors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maryann W Campion, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-48456
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Genetic Counseling Profession
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator analyzing the data will be blinded to which study arm participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meditation - Headspace (Experimental): Participants in this arm will be asked to meditate daily for 10 minutes for 8 weeks. Meditation instruction will be provided by the commercially available app/website Headspace (provided to participants for free). Participants in this arm will have access to the other meditation arm once they finish the study.
  Interventions: Behavioral: Meditation
- Meditation - Respite (Experimental): Participants in this arm will be asked to meditate daily for 10 minutes for 8 weeks. Meditation instruction will be provided by Respite, a website created by the investigators for this study. Participants in this arm will have access to the other meditation arm once they finish the study.
  Interventions: Behavioral: Meditation
- Observational (No Intervention): Participants in this arm will not receive any intervention. Their only study activity will be taking online surveys. They will have access to the two meditation arms once they finish the study.

INTERVENTIONS:
Behavioral: Meditation — 10 minutes a day of meditation, done on your own time.
  Arms: Meditation - Headspace; Meditation - Respite

SUMMARY:
This study is designed to determine whether meditation is beneficial for genetic counselors and genetic counseling students. The main goal is to see if meditation can help with professional well-being (burnout for genetic counselors, stress for genetic counseling students). The investigators will also explore whether meditation has other benefits for the genetic counseling profession.

DETAILED DESCRIPTION:
The investigators will recruit 390-420 genetic counselors and 189-210 genetic counseling students. Participants will be randomized into one of three groups of roughly the same size: two meditation groups and an observational group. All three groups will fill out online surveys at several points in the study. The only thing the observational group will be asked to do is fill out these surveys. The meditation groups will be asked to meditate for 10 minutes a day for 8 weeks. Participants will be provided with an app or website that instructs them on how to meditate.

Outcome analyses will be done with an intention to treat approach. Outcomes will be assessed using linear regression with the outcome variable as the dependent variable and baseline outcome measure, baseline mindfulness, and treatment group as the independent variables. Secondary outcomes will be considered exploratory.

The study is funded by the Jane Engelberg Memorial Foundation

ELIGIBILITY:
Inclusion Criteria:

* Genetic counselors who provide direct clinical care
* Genetic counseling students
* Self-reported fluency in English

Exclusion Criteria:

* Living outside the US

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Burnout (genetic counselors) | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  The primary outcome for genetic counselors is burnout, measured with the Professional Fulfillment Inventory
Stress (genetic counseling students) | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  The primary outcome for genetic counseling students is stress, measured with the Perceived Stress Scale

SECONDARY OUTCOMES:
Other dimensions of professional well-being: Stress (genetic counselors only) | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Perceived Stress Scale
Other dimensions of professional well-being: Professional fulfillment (genetic counselors only) | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Professional Fulfillment Index
Other dimensions of professional well-being: Reactive distress | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Interpersonal Reactivity Index
Other dimensions of professional well-being: Resilience | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Connor-Davidson Resilience Scale-10
Determinants of counseling effectiveness: Cognitive empathy | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Interpersonal Reactivity Index
Determinants of counseling effectiveness: Affective empathy | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Interpersonal Reactivity Index
Determinants of counseling effectiveness: Working alliance | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Working Alliance Inventory
Determinants of counseling effectiveness: Empathic understanding | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Barrett-Lennard Relationship Inventory
Determinants of counseling effectiveness: Unconditional positive regard | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Barrett-Lennard Relationship Inventory
Determinants of counseling effectiveness: Non-judging | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Five-Facet Mindfulness Questionnaire
Determinants of counseling effectiveness: Non-reactivity | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Measured with the Five-Facet Mindfulness Questionnaire
Retention in clinical roles | Measured at the end of the intervention period, typically 8 weeks after starting the study.
  Retention in clinical roles, measured we will measure intention to reduce clinical load, using a custom item with a visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Caleshu, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silver J, Caleshu C, Casson-Parkin S, Ormond K. Mindfulness Among Genetic Counselors Is Associated with Increased Empathy and Work Engagement and Decreased Burnout and Compassion Fatigue. J Genet Couns. 2018 Sep;27(5):1175-1186. doi: 10.1007/s10897-018-0236-6. Epub 2018 Mar 4. PMID 29502147